CLINICAL TRIAL: NCT05369377
Title: Zanubrutinib and Eltrombopag as Second-line Treatment for Patients With Immune Thrombocytopenia: a Multicentre, Open-label,Randomised, Controlled, Phase 2 Trial
Brief Title: Zanubrutinib and Eltrombopag as Second-line Treatment in Adults With Primary Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Navy General Hospital, Beijing (Other); Beijing Aerospace General Hospital (Other); Qilu Hospital of Shandong University (Other); Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zan-Eltro-ITP
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Immune Thrombocytopenia
Keywords: BTK inhibitor; Thrombopoietin-receptor agonist
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — zanubrutinib; eltrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zanubrutinib and eltrombopag (Experimental): Zanubrutinib 80mg po qd 6 weeks and eltrombopag 50 mg qd for up to 6 weeks.
  Interventions: Drug: Zanubrutinib; Drug: Eltrombopag
- Eltrombopag monotherapy (Active Comparator): Eltrombopag is given as 50 mg qd for up to 6 weeks.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib 80mg po qd 6 weeks
  Other Names: BTK inihibitor
  Arms: Zanubrutinib and eltrombopag
Drug: Eltrombopag — eltrombopag 50 mg qd for up to 6 weeks. The eltrombopag dose could be increased from 50 mg to 75 mg after 3 weeks in patients whose platelet counts were less than 50 000 per μL. Treatment was discontinued in patients who attained a platelet count greater than 200 000 per μL.

SUMMARY:
Randomized, open-label, multicenter study to compare the efficacy and safety of zanubrutinib plus eltrombopag compared to eltrombopag monotherapy for the first-line treatment of adults with chronic immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a prospective trial of patients with ITP in China. Zanubrutinib is administered as 80 mg po. qd for 6 weeks. Eltrombopag is given with 50 mg once daily for up to 6 weeks. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. This study assessed the efficacy and safety of eltrombopag plus zanubrutinib.

ELIGIBILITY:
Inclusion Criteria:

1. Primary immune thrombocytopenia (ITP) confirmed by excluding other supervened causes of thrombocytopenia;
2. Patients with chronic low platelet count (less than 30,000/µL) for 6 months who have failed at least one treatment for chronic low platelet count

2. Patients who did not achieve a sustained response to treatment with full-dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation 3. Willing and able to sign written informed consent

Exclusion Criteria:

1. Secondary immune thrombocytopenia (e.g., patients with HIV, HCV, Helicobacter pylori infection or patients with systemic lupus erythematosus)
2. congestive heart failure
3. severe arrhythmia
4. nursing or pregnant women
5. aspartate aminotransferase and alanine transaminase levels ≥ 3× the upper limit of the normal threshold criteria
6. creatinine or serum bilirubin levels each 1•5 times or more than the normal range
7. active or previous malignancy
8. Unable to do blood routine test for the sake of time, distance, economic issues or other reasons
9. History of clotting disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment response | 6 weeks
  The proportion of patients who had an increase in platelet counts to 50 000 per μL or more after 6 weeks of treatment

SECONDARY OUTCOMES:
Overall response | 6 weeks
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication after 6 weeks of treatment
Complete response (CR) | 6 weeks
  Complete response (CR) was defined as platelet count more than 100,000 per cubic millimeter and absence of bleeding
Time to response | 6 weeks
  The time from starting treatment to time of achievement of Response
Sustained response | 12 month
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 12-month follow-up
Number of patients with bleeding | 12 months
  Number of patients with bleeding complication ( WHO bleeding score)
Number of patients with adverse events | 12 months
  Number of patients with adverse events
Duration of response (DOR) | 12 months
  Duration of response at 12-month follow up
Loss of response | 12 months
  Platelet counts below 100 x 109/L or bleeding (from CR) or platelet counts below 30 x 109/L, less than 2-fold increase of baseline platelet count or bleeding (from R)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, md, Principal Investigator — Peking University People's Hospital, Peking University Insititute of Hematology
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided